CLINICAL TRIAL: NCT05055557
Title: The Role and Mechanism of O-GlcNAc Glycosylation Modified HAS2 in the Hyaluronic Acid Synthesis in ARDS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Southeast University, China (Other)
Responsible Party: Principal Investigator, Ling Liu, professor, Southeast University, China
Other Study IDs: ZDHMWHA
Record Dates: First submitted 2021-09-12; First posted 2021-09-24 (Actual); Last update posted 2021-09-24 (Actual); Status verified 2021-09

CONDITIONS: Hyaluronic Acid
Keywords: Acute respiratory distress syndrome; Pulmonary microvascular endothelial barrier;; Hyaluronic acid; Hyaluronic acid synthase 2
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Biospecimen Retention: Samples With DNA — whole blood samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- ARDS group: 1.85 years≥Age≥18 years. 2.Moderate-to-severe ARDS, defined by the ARDS Definition Task Force in the Berlin definition (partial pressure of arterial oxygen [PaO2]:FiO2 ratio ≤200 mmHg with a PEEP ≥5 cmH2O).
  3.Diagnosis of ARDS less than 72 hours. 4.Just observation
- Critically ill patients without ARDS group: Unstable vital signs, rapid changes in the condition, unstable function of more than two organ systems (excluding the respiratory system), decline or failure, the development of the disease may endanger the life of the patient.
- healthy adult group: Healthy adults, voluntarily join the study.

SUMMARY:
Maintaining the normal function of the pulmonary microvascular barrier is critical for ARDS treatment. To assess the relationship between the HAS2 protein level, HA content and the clinical prognosis of ARDS in patients with ARDS. Compare the HAS2 protein levels, HMW-HA and LMW-HA levels, endothelial injury indicators, and lungs in the blood of severe and non-ARDS severe patients and healthy adults admitted to the ICU. The correlation between permeability, disease severity and prognosis to explore the predictability of HAS2-HA on the clinical outcome of ARDS.

ELIGIBILITY:
Inclusion Criteria:

1.85 years≥Age≥18 years. 2.Moderate-to-severe ARDS, defined by the ARDS Definition Task Force in the Berlin definition (partial pressure of arterial oxygen [PaO2]:FiO2 ratio ≤200 mmHg with a PEEP ≥5 cmH2O).

3.Diagnosis of ARDS less than 72 hours.

Exclusion Criteria:

All patients who meet any of the following criteria will be excluded at enrollment and randomization.

1. Severe chronic respiratory diseases requiring long-term home oxygen therapy or noninvasive MV.
2. Undrained pneumothorax or subcutaneous emphysema.
3. Severe neuromuscular disease.
4. Hemodynamic instability (>30% increase in vasopressors within 6 hours or norepinephrine >0.5 ug/kg/min) (Am J Respir Crit Care Med. 2020; 201(2):178-187) .
5. Contraindications to hypercapnia, such as intracranial hypertension or acute coronary syndrome.
6. Severe other organs dysfunction with a low expected survival (7 days) or palliative care.
7. Solid organ or hematologic tumors with the expected survival time less than 30 days.
8. Participating in other clinical trials within 30 days.
9. Pregnancy.
10. Refusal to sign the informed consent.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1.85 years≥Age≥18 years. 2.Moderate-to-severe ARDS, defined by the ARDS Definition Task Force in the Berlin definition (partial pressure of arterial oxygen [PaO2]:FiO2 ratio ≤200 mmHg with a PEEP ≥5 cmH2O).
  3.Diagnosis of ARDS less than 72 hours.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-10-01 (Estimated); Primary Completion 2022-07-31 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
28-day fatality Rate | 28 days after enrollment
  28-day mortality (patients will be followed for 28 days)
90-day fatality rate | 90 days after enrollment
  90-day mortality (patients will be followed for 90 days)
ICU hospital stay | through study completion, an average of 4 week
  Length of ICU stay
ICU fatality rate | through study completion, an average of 4 week
  The ratio of the total number of deaths from all causes of the enrolled patients during ICU hospitalization.
Wearing time from mechanical ventilation | through study completion，an average of 4 week
  successful weaning defined as the absence of the requirement for ventilatory support, without reintubation
Peripheral blood HMW-HA and LMW-HA levels | 0, 1, 3, 7 days after enrollment
  ELISA method to separate and detect HMW-HA and LMW-HA levels（Units of Measure unit nM/ml）
HAS2 protein content in peripheral blood | 0, 1, 3, 7 days after enrollment
  ELISA method detects HAS2 protein in peripheral blood

SECONDARY OUTCOMES:
ENOS, ET-1, vWF levels in peripheral blood | 0, 1, 3, 7 days after enrollment
  ELISA method to detect eNOS, ET-1, vWF in peripheral blood to evaluate endothelial cell damage（Measure unit ng/ml）
Levels of bound mucinoglycans-1, nitric oxide, and acetylheparin sulfate in peripheral blood | 0, 1, 3, 7 days after enrollment
  glycocalyx levels of the endothelium were assessed by measuring the levels of mucin polysaccharide-1, nitric oxide and acetyl heparan sulfate in peripheral blood by ELISA assay（Measure unit ng/ml）
In peripheral blood, IL-1α, IL-6, neutrophils, lymphocytes, descending Procalcin, C-reactive protein value | 0, 1, 3, 7 days after enrollment
  The ELISA method detects IL-1α and IL-6 in the blood, and records the blood neutrophils, lymphocytes, and vary in procalcin and C-reactive protein to assess the inflammatory response of ARDS(Measure unit pg/ml）

IPD SHARING:
Plan to Share IPD: No